CLINICAL TRIAL: NCT05685264
Title: A PHASE 1, OPEN-LABEL, SINGLE DOSE STUDY TO INVESTIGATE THE PHARMACOKINETICS, PHARMACODYNAMICS, SAFETY, AND TOLERABILITY OF PONSEGROMAB ADMINISTERED SUBCUTANEOUSLY IN HEALTHY ADULT CHINESE PARTICIPANTS
Brief Title: A Study to Learn How the Study Medicine (Ponsegromab) is Changed and Eliminated From Healthy Chinese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C3651012
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Ponsegromab; Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ponsegromab low dose (Experimental)
  Interventions: Drug: Ponsegromab
- Ponsegromab high dose (Experimental)
  Interventions: Drug: Ponsegromab

INTERVENTIONS:
Drug: Ponsegromab — Participants will receive one subcutaneous injection
  Arms: Ponsegromab low dose
Drug: Ponsegromab — Participants will receive four subcutaneous injections
  Arms: Ponsegromab high dose

SUMMARY:
The purpose of this clinical trial is to learn about the safety of the study medicine (ponsegromab) and how it undergoes change and elimination in healthy Chinese adults. This study is seeking male and female Chinese participants who are very healthy as confirmed after some medical tests.

All participants in this study will receive Ponsegromab only once:

* for half of the participants, ponsegromab will be given as a shot in the front of the thigh, abdomen, or outer area of the upper arm at the study clinic.
* for another half of the participants, ponsegromab will be given as four shots in the front of the thigh, abdomen, or outer area of the upper arm at the study clinic.

We will measure the amount of the study medicine in the blood of the participants after giving the shots. Later we will examine experiences of people receiving the study medicine. This will help us understand how the medicine is changed and eliminated from your body and to decide if the study medicine is safe. Participants will take part in this study for 22 weeks. During this time, they will stay at the study clinic for the first 8 days and will visit the study clinic about 8 times.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 to 55 years of age, inclusive, at the time of signing the informed consent
2. Male and female Chinese participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, BP and PR measurement, 12-lead ECG, and laboratory tests. Chinese participants are defined as individuals currently residing in mainland China who were born in China and have both parents of Chinese descent.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
5. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Informed Consent Document..

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. History of HIV infection, syphilis, hepatitis B, or hepatitis C; positive testing for HIV, syphilis, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
3. History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody or molecules made of components of monoclonal antibodies.
4. History of recurrent infections or active infection within 28 days of screening.
5. History of sensitivity to heparin or heparin-induced thrombocytopenia.
6. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic (eg, contact with positive case, residence, or travel to an area with high incidence) that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
7. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
8. Exposure to live vaccines within 28 days of screening.
9. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or marketed or investigational monoclonal antibodies within 3 months or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
10. A positive urine drug test.
11. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
12. Screening 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTcF interval >450 msec, or QRS interval >120 msec). If the baseline uncorrected QT interval is >450 msec, this interval should be rate-corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
13. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * AST or ALT level ≥1.5 × ULN;
    * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
14. COVID-19 positive.
15. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 240 mL beer, 30 mL of 40% spirit or 90 mL of wine).
16. Blood donation (excluding plasma donations) of approximately 400 mL or more within 60 days prior to dosing.
17. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
18. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- China (2):
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - HuaShan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3651012

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 18 participants were screened and assigned to receive the study intervention. All of them received ponsegromab. All 18 participants completed treatment and follow-up phases.
Groups:
- Cohort 1: Ponsegromab 100 mg: Participants in Cohort 1 (ponsegromab 100 mg cohort) received a single subcutaneous (SC) dose of ponsegromab 100 mg on Day 1.
- Cohort 2: Ponsegromab 400 mg: Participants in Cohort 2 (ponsegromab 400 mg cohort) received a single SC dose of ponsegromab 400 mg on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: Ponsegromab 100 mg | Cohort 2: Ponsegromab 400 mg
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study intervention.
Groups:
- Cohort 1: Ponsegromab 100 mg: Participants in Cohort 1 (ponsegromab 100 mg cohort) received a single SC dose of ponsegromab 100 mg on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Ponsegromab 100 mg | Cohort 2: Ponsegromab 400 mg | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Median (Full Range); unit: Years] | 34.0 [27 to 54] | 25.0 [21 to 51] | 30.0 [21 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 9 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serum Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of Unbound and Total Ponsegromab
Description: AUCinf was defined as area under the serum concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: Pre-dose, 12, 24, 48, 72, 120, 168 hours after dose on Day 1, Days 10, 15, 29, 50, 71, 93, 106, and 127
Population: All enrolled participants who received a dose of ponsegromab and who had at least 1 of the serum pharmacokinetic (PK) parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)*day/milliliter (mL)
Arm/Group | Cohort 1: Ponsegromab 100 mg | Cohort 2: Ponsegromab 400 mg
Number analyzed (Participants) | 9 | 9
nanogram (ng)*day/milliliter (mL)
  Unbound ponsegromab: number analyzed (Participants) | 7 | 7
  Unbound ponsegromab | 109000 (58) | 590200 (59)
  Total ponsegromab | 350300 (21) | 1105000 (44)

2. Primary Outcome: Area Under the Serum Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Unbound and Total Ponsegromab
Description: AUClast was defined as area under the serum concentration-time profile from time 0 to the time of the last quantifiable concentration.
Time Frame: Pre-dose, 12, 24, 48, 72, 120, 168 hours after dose on Day 1, Days 10, 15, 29, 50, 71, 93, 106, and 127
Population: All enrolled participants who received a dose of ponsegromab and who had at least 1 of the serum PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*day/mL
Arm/Group | Cohort 1: Ponsegromab 100 mg | Cohort 2: Ponsegromab 400 mg
Number analyzed (Participants) | 9 | 9
ng*day/mL
  Unbound ponsegromab | 95170 (55) | 647700 (60)
  Total ponsegromab | 337800 (20) | 1036000 (42)

3. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Unbound and Total Ponsegromab
Description: Cmax was defined as maximum observed concentration. Cmax was observed directly from data.
Time Frame: Pre-dose, 12, 24, 48, 72, 120, 168 hours after dose on Day 1, Days 10, 15, 29, 50, 71, 93, 106, and 127
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: Ponsegromab 100 mg | Cohort 2: Ponsegromab 400 mg
Number analyzed (Participants) | 9 | 9
ng/mL
  Unbound ponsegromab | 4698 (41) | 21330 (64)
  Total ponsegromab | 6978 (28) | 24910 (60)

4. Primary Outcome: Time for Cmax (Tmax) of Unbound and Total Ponsegromab
Description: Tmax was defined as time for Cmax. Tmax was observed directly from data as time of first occurrence.
Time Frame: Pre-dose, 12, 24, 48, 72, 120, 168 hours after dose on Day 1, Days 10, 15, 29, 50, 71, 93, 106, and 127
Population: as for outcome 2
Measure: Median (Full Range); unit: day
Arm/Group | Cohort 1: Ponsegromab 100 mg | Cohort 2: Ponsegromab 400 mg
Number analyzed (Participants) | 9 | 9
day
  Unbound ponsegromab | 7.01 [5.00 to 14.0] | 5.00 [3.00 to 14.0]
  Total ponsegromab | 7.01 [3.00 to 14.0] | 6.99 [3.00 to 28.0]

5. Primary Outcome: Terminal Half Life (t1/2) of Unbound and Total Ponsegromab
Description: t1/2 was defined as terminal half life. t1/2 was calculated as Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log linear concentration time curve.
Time Frame: Pre-dose, 12, 24, 48, 72, 120, 168 hours after dose on Day 1, Days 10, 15, 29, 50, 71, 93, 106, and 127
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Cohort 1: Ponsegromab 100 mg | Cohort 2: Ponsegromab 400 mg
Number analyzed (Participants) | 9 | 9
day
  Unbound ponsegromab: number analyzed (Participants) | 7 | 7
  Unbound ponsegromab | 8.393 (2.8461) | 10.37 (3.7287)
  Total ponsegromab | 23.40 (3.8135) | 31.09 (8.9457)

6. Secondary Outcome: Number of Participants With All-Causality Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were defined as events that started on or after the first dose but before the end of the study (approximately 18 weeks post dose on Day 1). An SAE was defined as any untoward medical occurrence at any dose that resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect.
Time Frame: From the first dose of study intervention on Day 1 to Day 127
Population: All enrolled participants who received a dose of ponsegromab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ponsegromab 100 mg | Cohort 2: Ponsegromab 400 mg
Number analyzed (Participants) | 9 | 9
Participants
  TEAEs | 4 | 7
  SAEs | 0 | 0

7. Secondary Outcome: Number of Participants With Treatment-Related TEAEs and SAEs
Description: AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were defined as events that started on or after the first dose but before the end of the study (approximately 18 weeks post dose on Day 1). An SAE was defined as any untoward medical occurrence at any dose that resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect. Causality of the TEAEs and SAEs was judged by the investigator.
Time Frame: From the first dose of study intervention on Day 1 to Day 127
Population: All enrolled participants who received a dose of ponsegromab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ponsegromab 100 mg | Cohort 2: Ponsegromab 400 mg
Number analyzed (Participants) | 9 | 9
Participants
  TEAEs | 0 | 1
  SAEs | 0 | 0

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities Without Regard to Baseline Abnormality
Description: Hematology parameters included hemoglobin, hematocrit, red blood cell, white blood cell and platelet count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, mean platelet volume, total neutrophils, eosinophils, monocytes, basophils and lymphocytes. Chemistry parameters included blood urea nitrogen, glucose (fasting), calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein, and creatinine. Urine parameters included pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, microscopy. Only those categories in which at least 1 participant had data were reported.
Time Frame: From the first dose of study intervention on Day 1 to Day 127
Population: All enrolled participants who received a dose of ponsegromab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ponsegromab 100 mg | Cohort 2: Ponsegromab 400 mg
Number analyzed (Participants) | 9 | 9
Participants
  Ery. Mean Corpuscular HGB Concentration (g/dL) >1.1 x upper limit of normal (ULN) | 0 | 1
  Mean Platelet Volume (fL) <0.9 x lower limit of normal (LLN) | 4 | 2
  Lymphocytes (10^3/mm^3) >1.2 x ULN | 0 | 1
  Neutrophils (10^9/L) <0.8 x LLN | 0 | 1
  Alanine Aminotransferase (U/L) >3.0 x ULN | 0 | 1
  Urate (mg/dL) >1.2 x ULN | 1 | 1
  pH (Scalar) <1.0 x LLN | 6 | 5
  Ketones ≥1 | 1 | 5
  Urine Hemoglobin ≥1 | 1 | 1
  Urobilinogen ≥1 | 0 | 3
  Leukocyte Esterase ≥1 | 2 | 3
  Urine Leukocytes (/uL) >1.0 x ULN | 1 | 1
  Epithelial Cells ≥6 | 1 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Change in Vital Signs
Description: Vital sign measurements included supine blood pressure and pulse rate. Any safety assessments (vital sign measurements) including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator or were considered meeting the AE definition and are listed below.
Time Frame: From the first dose of study intervention on Day 1 to Day 127
Population: All enrolled participants who received a dose of ponsegromab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ponsegromab 100 mg | Cohort 2: Ponsegromab 400 mg
Number analyzed (Participants) | 9 | 9
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Change in Electrocardiogram (ECG)
Description: ECG abnormalities criteria included: 1) maximum QTc interval adjusted according to Fridericia formula (QTcF) (msec): >450, >480, >500, increase from baseline >30, increase from baseline >30, >60; 2) maximum pulse rate (msec): ≥300, baseline >200 and maximum increase ≥25%, baseline ≤200 and maximum increase ≥50%; 3) maximum QRS (msec): ≥140, increase ≥50%.
Time Frame: From the first dose of study intervention on Day 1 to Day 127
Population: All enrolled participants who received a dose of ponsegromab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ponsegromab 100 mg | Cohort 2: Ponsegromab 400 mg
Number analyzed (Participants) | 9 | 9
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study intervention on Day 1 to Day 127
Arm/Group | Cohort 1: Ponsegromab 100 mg | Cohort 2: Ponsegromab 400 mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 4/9 | 7/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ponsegromab 100 mg (N=9) | Cohort 2: Ponsegromab 400 mg (N=9)
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 2
Gingivitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Urine ketone body present (Investigations) | 0 | 1
Urine leukocyte esterase positive (Investigations) | 0 | 2
Urobilinogen urine increased (Investigations) | 0 | 1
White blood cells urine positive (Investigations) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT05685264/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT05685264/SAP_001.pdf